CLINICAL TRIAL: NCT04709107
Title: Validation of Electronic Version of the VascuQoL-6 Questionnaire to Assess Patient Related Outcome Measures (ePROM) After Revascularization for Lower Limb Peripheral Arterial Disease in German-speaking Part of Switzerland
Brief Title: Validation of the VascuQoL-6 Questionnaire to Assess ePROM After Revascularization for Lower Limb Peripheral Arterial Disease in German-speaking Part of Switzerland
Acronym: VascuQol6ValCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Andrej Isaak, Head of Vascular Surgery, Kantonsspital Aarau
Other Study IDs: 2020-00689
Record Dates: First submitted 2020-12-28; First posted 2021-01-14 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease, pad, quality of life, ePROM, patient related outcome measures, HRQoL, health related quality of life
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elective: Patients undergoing elective revascularisation (endovascular or surgical) for PAD.
  Interventions: Other: Quality of life assessment - elective
- Emergent: Patients undergoing emergent revascularisation (endovascular or surgical) for PAD.
  Interventions: Other: Quality of life assessment - emergent

INTERVENTIONS:
Other: Quality of life assessment - elective — Patients will be asked to fill up both VascuQoL-6 and SF-36 questionnaires before the procedure, as well at 30-days and 1-year follow-up visit while they are sitting in the waiting room. To assess reliability and systematic shift and variation between the two assessments, elective patients will be asked to fill the VascuQoL-6 again at the admission to hospital, as well as 1 week after the 30-days follow-up vie an e-mail link for a test-retest assessment. All questionnaires will be administered on a tablet.
  During the 30-days follow-up 4 extra questions concerning patient related outcomes and occurrence of major complication will be added to the VascuQoL-6 questionnaire in the App. During every visit (preoperatively, at 30-days and 1-year follow-up) the stage of the lower limb peripheral artery disease will be noted according to the WIfI-Classification.
  Groups: Elective
Other: Quality of life assessment - emergent — Patients will be asked to fill up both VascuQoL-6 and SF-36 questionnaires before the procedure, as well at 30-days and 1-year follow-up visit while they are sitting in the waiting room. All questionnaires will be administered on a tablet.
  During the 30-days follow-up 4 extra questions concerning patient related outcomes and occurrence of major complication will be added to the VascuQoL-6 questionnaire in the App. During every visit (preoperatively, at 30-days and 1-year follow-up) the stage of the lower limb peripheral artery disease will be noted according to the WIfI-Classification.
  Groups: Emergent

SUMMARY:
Two hundred patients evaluated to undergo revascularization (elective/emergent, surgical/interventional) for lower limb PAD at the cantonal hospital of Aarau, Switzerland, will, after consenting to participate in the study, be asked to fill up both SF-36 and VascuQol-6 questionnaires while sitting in a waiting room before the procedure and during the 30 days and 1-year routine follow up. An electronic version of the questionnaires will be administered on a tablet. The primary goal is to validate the clinical use of the German electronic version of the VascuQol-6 questionnaire to assess patient-related outcomes of the performed treatment by patients with PAD.

DETAILED DESCRIPTION:
Lower extremity peripheral artery disease is a chronic illness that has a significant effect on the quality of life of the patients in short- as well as long-term.

Generic Instruments, such as widely used Medical Outcomes Study Short Form 36 questionnaire (SF-36) might be too insensitive to specific problems and associated comorbidities of vascular surgery patients as well as too complicated for routine use in a busy clinical setting. Therefore, the Vascular Quality of life questionnaire (VascuQoL-25) has been developed for use in the UK in 2001 at the Vascular Surgical Unit of King's College Hospital in London. To further simplify the use of the questionnaire, a lighter Version, that reduced the amount of asked questions from 25 to 6 (VascQuol-6) has been presented and found to be both valid and relevant. VascuQoL- 6 is a disease-specific questionnaire, developed to assess health-related quality of life (HRQoL) in patients with peripheral artery disease. It has been translated to 8 languages including German, and successfully validated for the use to assess in patients with peripheral artery disease in Sweden, Netherlands, Norway, Brazil and Poland.

In opinion of the investigators, a unified means to obtain relevant data concerning patient-related outcomes following treatment (endovascular or surgical) for PAD as part of existing aftercare schemes currently lacks in Switzerland. A simple tool such as VascuQoL-6 would allow collecting and objectively assessing, as well as comparing this kind of information after such procedures.

The main objective of the project is to validate the electronic version of the VascuQoL-6 for assessment of patient-related outcomes after a revascularization procedure (either surgical or interventional) for peripheral artery disease in the German-speaking part of Switzerland preoperatively, during the routine 30 days and a one-year follow-up.

Furthermore, upon the successful validation of the electronic VascuQoL-6, the investigators seek to implement the use of this easy to use, straight-forward tool in the follow-up scheme of the Swiss Vascular Registry (SwissVasc).

This project is of Risk A (minimum risk) according to art. 7 (HRO), because the patient-related quality of life will be evaluated after vascular surgery or intervention and will not have an influence on treatment modality.

Hypothesis and primary objective Assessment of quality regarding invasive treatment (endovascular or surgical), outcomes and patients satisfaction becomes a more and more powerful instrument to influence and guide decisions in the Swiss healthcare system. However, no unified means are currently being applied as part of the existing follow-up schema after revascularization for PAD in the German-speaking part of Switzerland. Therefore, the possibility to provide, assess, compare and use the information about short- mid- and long-term patient-related outcomes and improved/decreased disease- related quality of life in the decision-making process is limited.

Validation of a comprehensible and easy-to-use electronic Version of the VascuQoL-6 will allow obtaining such information in patients that underwent vascular/ endovascular surgery in the German-speaking part of Switzerland.

SwissVasc (i.e. Adjumed.net) is a nation-wide database to register vascular interventions and associated outcomes. Registration of individual data in SwissVasc (i.e. 30-day mortality, complication rate) is mandatory in Kanton Zurich and will become mandatory in Kanton Basel- Stadt and Basel-Landschaft in 2020. Moreover, this register will soon be part of the statutes of the Swiss Society of Vascular Surgery to evaluate the quality of training in each institution.

The Evaluation of VascuQoL-6 is part of this ambitious project. The goal is to implement the use of this questionnaire into the SwissVasc registry follow-up schema, to provide a uniformly used tool to collect and investigate the above-said information.

ELIGIBILITY:
Inclusion Criteria:

* confirmed PAD
* elective or emergent revascularization indicated (surgery/intervention)
* native German speakers - no cognitive impairment

Exclusion Criteria:

* not fulfilling any of the inclusion criteria
* patients refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteer native German-speakers with no cognitive impairment, by whom an elective or emergent revascularisation (endovascular or surgical) for lower limb peripheral artery disease has been indicated.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
VascuQoL-6 Score | baseline
  Disease specific Questionnaire for peripheral arterial Disease, consists of 6 questions
VascuQoL-6 Score | 1 Month after revascularisation
  Disease specific Questionnaire for peripheral arterial Disease, consists of 6 questions
VascuQoL-6 Score | 1 year after revascularisation
  Disease specific Questionnaire for peripheral arterial Disease, consists of 6 questions

SECONDARY OUTCOMES:
WIfl classification | baseline
  Wound, Ischemia and foot Infection Classification system - used to predict 1-year amputation risk and potential benefit of revascularization. The wound, limb Ischemia and foot infection are stratified and graded, thus creating a score.
WIfl classification | 1 month after revascularisation
  Wound, Ischemia and foot Infection Classification system - used to predict 1-year amputation risk and potential benefit of revascularization. The wound, limb Ischemia and foot infection are stratified and graded, thus creating a score.
WIfl classification | 1 year after revascularisation
  Wound, Ischemia and foot Infection Classification system - used to predict 1-year amputation risk and potential benefit of revascularization. The wound, limb Ischemia and foot infection are stratified and graded, thus creating a score.
Complication rates | 1 year
  Occurence of myocardial infarction, stroke or death
Ankle-brachial indices | baseline
  Ankle pressure to brachial pressure index, used to evaluate PAD
Ankle-brachial indices | 1 month after revascularisation
  Ankle pressure to brachial pressure index, used to evaluate PAD
Ankle-brachial indices | 1 year after revascularisation
  Ankle pressure to brachial pressure index, used to evaluate PAD
Puls-plethysmography | baseline
  Plethysmography is routine examination for PAD, allows for evaluation of extremity perfusion at different levels
Puls-plethysmography | 1 month after revascularisation
  Plethysmography is routine examination for PAD, allows for evaluation of extremity perfusion at different levels
Puls-plethysmography | 1 year after revascularisation
  Plethysmography is routine examination for PAD, allows for evaluation of extremity perfusion at different levels
SF-36 Score | baseline
  Short Form 36 Questionnaire - acknowledged tool for assesment of health related quality of life. Not disease specific, used as gold standard to evaluate the VascuQol-6 Questionnaire
SF-36 Score | 1 month after revascularisation
  Short Form 36 Questionnaire - acknowledged tool for assesment of health related quality of life. Not disease specific, used as gold standard to evaluate the VascuQol-6 Questionnaire
SF-36 Score | 1 year after revascularisation
  Short Form 36 Questionnaire - acknowledged tool for assesment of health related quality of life. Not disease specific, used as gold standard to evaluate the VascuQol-6 Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Isaak, Dr. med., Study Director — Kantonsspital Aarau
Locations (1):
- Kantonsspital Aarau, Aarau, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Morgan MB, Crayford T, Murrin B, Fraser SC. Developing the Vascular Quality of Life Questionnaire: a new disease-specific quality of life measure for use in lower limb ischemia. J Vasc Surg. 2001 Apr;33(4):679-87. doi: 10.1067/mva.2001.112326. PMID 11296317
- [Background] Nordanstig J, Wann-Hansson C, Karlsson J, Lundstrom M, Pettersson M, Morgan MB. Vascular Quality of Life Questionnaire-6 facilitates health-related quality of life assessment in peripheral arterial disease. J Vasc Surg. 2014 Mar;59(3):700-7. doi: 10.1016/j.jvs.2013.08.099. Epub 2013 Dec 15. PMID 24342060
- [Background] Conway K, et al. Linguistic validation of the vascular quality of life questionnaire (VASCUQOL) in 8 languages. Value in Health. 2000, 3(2):113.
- [Background] Kumlien C, Nordanstig J, Lundstrom M, Pettersson M. Validity and test retest reliability of the vascular quality of life Questionnaire-6: a short form of a disease-specific health-related quality of life instrument for patients with peripheral arterial disease. Health Qual Life Outcomes. 2017 Sep 29;15(1):187. doi: 10.1186/s12955-017-0762-1. PMID 28962624
- [Background] Larsen ASF, Reiersen AT, Jacobsen MB, Klow NE, Nordanstig J, Morgan M, Wesche J. Validation of the Vascular quality of life questionnaire - 6 for clinical use in patients with lower limb peripheral arterial disease. Health Qual Life Outcomes. 2017 Sep 22;15(1):184. doi: 10.1186/s12955-017-0760-3. PMID 28938901
- [Background] de Almeida Correia M, Andrade-Lima A, Mesquita de Oliveira PL, Domiciano RM, Ribeiro Domingues WJ, Wolosker N, Puench-Leao P, Ritti-Dias RM, Cucato GG. Translation and Validation of the Brazilian-Portuguese Short Version of Vascular Quality of Life Questionnaire in Peripheral Artery Disease Patients with Intermittent Claudication Symptoms. Ann Vasc Surg. 2018 Aug;51:48-54.e1. doi: 10.1016/j.avsg.2018.02.026. Epub 2018 May 15. PMID 29772330
- [Background] Belowski A, Partyka L, Krzanowski M, Polczyk R, Maga P, Maga M, Acquadro C, Lambe J, Morgan M, Nizankowski R. Clinical and linguistic validation of the Polish version of VascuQol: a disease-specific quality-of-life questionnaire assessing patients with chronic limb ischemia. Pol Arch Intern Med. 2019 Mar 29;129(3):167-174. doi: 10.20452/pamw.4455. Epub 2019 Feb 22. PMID 30793704
- [Background] Conte MS, Bradbury AW, Kolh P, White JV, Dick F, Fitridge R, Mills JL, Ricco JB, Suresh KR, Murad MH, Aboyans V, Aksoy M, Alexandrescu VA, Armstrong D, Azuma N, Belch J, Bergoeing M, Bjorck M, Chakfe N, Cheng S, Dawson J, Debus ES, Dueck A, Duval S, Eckstein HH, Ferraresi R, Gambhir R, Gargiulo M, Geraghty P, Goode S, Gray B, Guo W, Gupta PC, Hinchliffe R, Jetty P, Komori K, Lavery L, Liang W, Lookstein R, Menard M, Misra S, Miyata T, Moneta G, Munoa Prado JA, Munoz A, Paolini JE, Patel M, Pomposelli F, Powell R, Robless P, Rogers L, Schanzer A, Schneider P, Taylor S, De Ceniga MV, Veller M, Vermassen F, Wang J, Wang S; GVG Writing Group for the Joint Guidelines of the Society for Vascular Surgery (SVS), European Society for Vascular Surgery (ESVS), and World Federation of Vascular Societies (WFVS). Global Vascular Guidelines on the Management of Chronic Limb-Threatening Ischemia. Eur J Vasc Endovasc Surg. 2019 Jul;58(1S):S1-S109.e33. doi: 10.1016/j.ejvs.2019.05.006. Epub 2019 Jun 8. PMID 31182334
- [Background] Cull DL, Manos G, Hartley MC, Taylor SM, Langan EM, Eidt JF, Johnson BL. An early validation of the Society for Vascular Surgery lower extremity threatened limb classification system. J Vasc Surg. 2014 Dec;60(6):1535-41. doi: 10.1016/j.jvs.2014.08.107. Epub 2014 Oct 3. PMID 25282695
- [Background] Zhan LX, Branco BC, Armstrong DG, Mills JL Sr. The Society for Vascular Surgery lower extremity threatened limb classification system based on Wound, Ischemia, and foot Infection (WIfI) correlates with risk of major amputation and time to wound healing. J Vasc Surg. 2015 Apr;61(4):939-44. doi: 10.1016/j.jvs.2014.11.045. Epub 2015 Feb 2. PMID 25656592